CLINICAL TRIAL: NCT03940248
Title: Phase II Study to Evaluate the Cosmetic Outcome of Using Pencil Beam Scanning Proton Therapy for Accelerated Partial Breast Irradiation in Early Stage Breast Cancer
Brief Title: Proton Accelerated Partial Breast Irradiation
Acronym: APBI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to insurance non-payment, no subjects were enrolled.
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Teresa Meier, Associate Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0088
Record Dates: First submitted 2019-04-22; First posted 2019-05-07 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: Proton Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Stage Breast Cancer (Experimental): Patients to be treated with Accelerated Partial Breast Irradiation utilizing pencil beam scanning proton therapy. Treatment will be delivered twice a day, at least 6 hours apart, over 5 treatment days.
  Interventions: Radiation: Proton Accelerated Partial Breast Irradiation

INTERVENTIONS:
Radiation: Proton Accelerated Partial Breast Irradiation — 38.5 Cobalt Gray Equivalent (CGE) given over 10 fractions

SUMMARY:
This prospective, non-randomized phase II study will evaluate the cosmetic outcome of using pencil beam scanning proton therapy for partial breast irradiation in patients diagnosed with early stage breast cancer. In addition the study will evaluate the acute and late toxicities, and the rates of ipsilateral breast tumor recurrence, both in situ and invasive disease.

To qualify for the trial, patients must be 50 years or older and have stage 0 (carcinoma in situ) or stage IA or IIA invasive carcinoma of the breast with no evidence of metastatic disease. The tumor size must be 3cm or less. Women must have undergone a partial mastectomy with margins free of invasive cancer and at least a 2mm margin for in situ disease. Patients must have clinically node negative disease. Patients with invasive disease must also have nodal assessment performed with either sentinel lymph node biopsy or axillary lymph node dissection and patients must have pathologically node negative disease. Accelerated partial breast irradiation (APBI) will utilize pencil beam scanning proton therapy. Partial breast irradiation will be delivered twice a day, at least 6 hours apart, over 5 treatment days.

This trial is designed to accrue 21 patients over a period of three years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must consent to be in the study and must have signed an approved consent form conforming with institutional guidelines.
* Patients must be ≥ 50 years old.
* Patients should have a life expectancy of at least 10 years taking into consideration comorbid conditions.
* Surgical treatment of the breast must have been partial mastectomy. The margins of the resected specimen must be histologically free of tumor for invasive disease and with at least a 2mm margin for in situ disease. Reexcision of surgical margins is permitted to obtain negative margins. Postoperative mammogram of the surgical specimen or breast must be performed to confirm that all abnormal calcifications were removed at the time of surgery. Surgical clips must be placed at the partial mastectomy site by the surgeon at the time of excision.
* Patients must have American Joint Committee on Cancer 8th edition pathology stage Tis, T1, or T2 and N0 as assessed by sentinel lymph node biopsy or axillary lymph node dissection for invasive disease. The tumor size must be 3cm or less in greatest dimension.
* On histologic examination, the tumor must be ductal carcinoma in situ (low or intermediate grade), invasive ductal carcinoma (any grade), or invasive lobular carcinoma.
* Patients must have unicentric disease with limited or focal lymphovascular space invasion (LVSI).
* Patients must have an estrogen reception (ER) analysis performed and the primary tumor should be ER positive.
* The target partial mastectomy cavity must be clearly delineated and the target partial mastectomy cavity/whole breast reference volume must be ≤ 30% based on the post- operative scan. The partial mastectomy cavity must be > 5mm from the skin. This can be confirmed at time of CT simulation for radiation treatment planning.
* Patients must enroll within 42 days following the last surgery for breast cancer (partial mastectomy or re-excision of margins).
* Proton APBI should start within 12 weeks from the time of surgery.

Exclusion Criteria:

* Male
* Patients < 50 years of age.
* Tumor > 3cm in greatest dimension or American Joint Committee on Cancer 8th edition pathologic stage T3 or T4 or node positive disease.
* If patients have invasive carcinoma and no nodal assessment was performed, specifically the patient did not undergo sentinel lymph node biopsy or axillary lymph node dissection.
* Patients with persistently positive margins despite attempted re-excision.
* Proven multicentric disease or extensive LVSI.
* Clear delineation of the extent of the target partial mastectomy cavity is not possible.
* Patients who have undergone oncoplastic reconstruction.
* Any patients who received neoadjuvant chemotherapy or hormonal therapy prior to surgical excision of the tumor.
* Any patients who require adjuvant chemotherapy following lumpectomy.
* Patients whose primary tumor is ER negative.
* Patients with high grade ductal carcinoma in situ.
* Patients with known BRCA1 or BRCA2 mutation.
* Prior breast or thoracic radiation and any prior breast surgery in the ipsilateral breast.
* Patients with history of collagen vascular disease including scleroderma, lupus, polymyositis, or dermatomyositis.
* Pregnancy.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Cosmetic outcome (change in appearance as compared to untreated breast) | Through Study Completion, an average of 2 years
  Breast Cancer Treatment Outcome Scale [8 (no difference) through 32 (large difference)]
Cosmetic outcome (change in appearance as compared to untreated breast) | Through Study Completion, an average of 2 years
  Physician and Nurse Harvard Cosmesis Scale [1 (excellent) through 4 (poor)]

SECONDARY OUTCOMES:
Rates of acute (within 3 months of treatment) toxicity | Through Study Completion, an average of 2 years
  Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Rates of late (> 3 months after treatment) toxicity | Through Study Completion, an average of 2 years
  Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Rate of ipsilateral breast tumor recurrence, including both in situ and invasive disease. | Through Study Completion, an average of 2 years
  Presence of invasive or ductal carcinoma in-situ in ipsilateral breast as confirmed by biopsy
Rate of regional recurrence | Through Study Completion, an average of 2 years
  Presence of tumor in the ipsilateral axillary, infraclavicular, supraclavicular or internal mammary lymph nodes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howlader N, N.A., Krapcho M, Miller D, Bishop K, Kosary CL, Yu M, Ruhl J, Tatalovich Z, Mariotto A, Lewis DR, Chen HS, Feuer EJ, Cronin KA (eds). . SEER Cancer Statistics Review, 1975-2014, National Cancer Institute. . 2017; Available from: https://seer.cancer.gov/csr/1975_2014/
- [Background] van Dongen JA, Voogd AC, Fentiman IS, Legrand C, Sylvester RJ, Tong D, van der Schueren E, Helle PA, van Zijl K, Bartelink H. Long-term results of a randomized trial comparing breast-conserving therapy with mastectomy: European Organization for Research and Treatment of Cancer 10801 trial. J Natl Cancer Inst. 2000 Jul 19;92(14):1143-50. doi: 10.1093/jnci/92.14.1143. PMID 10904087
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Byun, D.J., et al., Omission of Adjuvant Radiation Therapy Following Breast Conservation Surgery for Ductal Carcinoma In Situ: Analysis of the National Cancer Data Base. International Journal of Radiation Oncology • Biology • Physics. 96(2): p. E38.
- [Background] Feigelson HS, Carroll NM, Weinmann S, Haque R, Yu CL, Butler MG, Waitzfelder B, Wrenn MG, Capra A, McGlynn EA, Habel LA. Treatment patterns for ductal carcinoma in situ from 2000-2010 across six integrated health plans. Springerplus. 2015 Jan 17;4:24. doi: 10.1186/s40064-014-0776-7. eCollection 2015. PMID 25625043
- [Background] Fisher J, Scott C, Stevens R, Marconi B, Champion L, Freedman GM, Asrari F, Pilepich MV, Gagnon JD, Wong G. Randomized phase III study comparing Best Supportive Care to Biafine as a prophylactic agent for radiation-induced skin toxicity for women undergoing breast irradiation: Radiation Therapy Oncology Group (RTOG) 97-13. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1307-10. doi: 10.1016/s0360-3016(00)00782-3. PMID 11121627
- [Background] Fernando IN, Ford HT, Powles TJ, Ashley S, Glees JP, Torr M, Grafton D, Harmer CL. Factors affecting acute skin toxicity in patients having breast irradiation after conservative surgery: a prospective study of treatment practice at the Royal Marsden Hospital. Clin Oncol (R Coll Radiol). 1996;8(4):226-33. doi: 10.1016/s0936-6555(05)80657-0. PMID 8871000
- [Background] Krauss DJ, Kestin LL, Mitchell C, Martinez AA, Vicini FA. Changes in temporal patterns of local failure after breast-conserving therapy and their prognostic implications. Int J Radiat Oncol Biol Phys. 2004 Nov 1;60(3):731-40. doi: 10.1016/j.ijrobp.2004.04.010. PMID 15465189
- [Background] Polgar C, Fodor J, Major T, Nemeth G, Lovey K, Orosz Z, Sulyok Z, Takacsi-Nagy Z, Kasler M. Breast-conserving treatment with partial or whole breast irradiation for low-risk invasive breast carcinoma--5-year results of a randomized trial. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):694-702. doi: 10.1016/j.ijrobp.2007.04.022. Epub 2007 May 25. PMID 17531400
- [Background] Vicini F, Winter K, Wong J, Pass H, Rabinovitch R, Chafe S, Arthur D, Petersen I, White J, McCormick B. Initial efficacy results of RTOG 0319: three-dimensional conformal radiation therapy (3D-CRT) confined to the region of the lumpectomy cavity for stage I/ II breast carcinoma. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):1120-7. doi: 10.1016/j.ijrobp.2009.06.067. Epub 2009 Nov 10. PMID 19910132
- [Background] Chafe S, Moughan J, McCormick B, Wong J, Pass H, Rabinovitch R, Arthur DW, Petersen I, White J, Vicini FA. Late toxicity and patient self-assessment of breast appearance/satisfaction on RTOG 0319: a phase 2 trial of 3-dimensional conformal radiation therapy-accelerated partial breast irradiation following lumpectomy for stages I and II breast cancer. Int J Radiat Oncol Biol Phys. 2013 Aug 1;86(5):854-9. doi: 10.1016/j.ijrobp.2013.04.005. Epub 2013 May 29. PMID 23726000
- [Background] Vaidya JS, Bulsara M, Wenz F, Coombs N, Singer J, Ebbs S, Massarut S, Saunders C, Douek M, Williams NR, Joseph D, Tobias JS, Baum M. Reduced Mortality With Partial-Breast Irradiation for Early Breast Cancer: A Meta-Analysis of Randomized Trials. Int J Radiat Oncol Biol Phys. 2016 Oct 1;96(2):259-265. doi: 10.1016/j.ijrobp.2016.05.008. Epub 2016 May 13. PMID 27478165
- [Background] Correa C, Harris EE, Leonardi MC, Smith BD, Taghian AG, Thompson AM, White J, Harris JR. Accelerated Partial Breast Irradiation: Executive summary for the update of an ASTRO Evidence-Based Consensus Statement. Pract Radiat Oncol. 2017 Mar-Apr;7(2):73-79. doi: 10.1016/j.prro.2016.09.007. Epub 2016 Sep 17. PMID 27866865
- [Background] Wang X, Amos RA, Zhang X, Taddei PJ, Woodward WA, Hoffman KE, Yu TK, Tereffe W, Oh J, Perkins GH, Salehpour M, Zhang SX, Sun TL, Gillin M, Buchholz TA, Strom EA. External-beam accelerated partial breast irradiation using multiple proton beam configurations. Int J Radiat Oncol Biol Phys. 2011 Aug 1;80(5):1464-72. doi: 10.1016/j.ijrobp.2010.04.052. Epub 2010 Aug 12. PMID 20708848
- [Background] Taghian AG, Kozak KR, Katz A, Adams J, Lu HM, Powell SN, DeLaney TF. Accelerated partial breast irradiation using proton beams: Initial dosimetric experience. Int J Radiat Oncol Biol Phys. 2006 Aug 1;65(5):1404-10. doi: 10.1016/j.ijrobp.2006.03.017. Epub 2006 May 26. PMID 16730137
- [Background] Wisenbaugh ES, Andrews PE, Ferrigni RG, Schild SE, Keole SR, Wong WW, Vora SA. Proton beam therapy for localized prostate cancer 101: basics, controversies, and facts. Rev Urol. 2014;16(2):67-75. PMID 25009446
- [Background] Hall EJ. Intensity-modulated radiation therapy, protons, and the risk of second cancers. Int J Radiat Oncol Biol Phys. 2006 May 1;65(1):1-7. doi: 10.1016/j.ijrobp.2006.01.027. PMID 16618572
- [Background] Bush DA, Slater JD, Garberoglio C, Do S, Lum S, Slater JM. Partial breast irradiation delivered with proton beam: results of a phase II trial. Clin Breast Cancer. 2011 Aug;11(4):241-5. doi: 10.1016/j.clbc.2011.03.023. Epub 2011 Jun 12. PMID 21729673
- [Background] Galland-Girodet S, Pashtan I, MacDonald SM, Ancukiewicz M, Hirsch AE, Kachnic LA, Specht M, Gadd M, Smith BL, Powell SN, Recht A, Taghian AG. Long-term cosmetic outcomes and toxicities of proton beam therapy compared with photon-based 3-dimensional conformal accelerated partial-breast irradiation: a phase 1 trial. Int J Radiat Oncol Biol Phys. 2014 Nov 1;90(3):493-500. doi: 10.1016/j.ijrobp.2014.04.008. Epub 2014 May 29. PMID 24880212
- [Background] Kozak KR, Smith BL, Adams J, Kornmehl E, Katz A, Gadd M, Specht M, Hughes K, Gioioso V, Lu HM, Braaten K, Recht A, Powell SN, DeLaney TF, Taghian AG. Accelerated partial-breast irradiation using proton beams: initial clinical experience. Int J Radiat Oncol Biol Phys. 2006 Nov 1;66(3):691-8. doi: 10.1016/j.ijrobp.2006.06.041. PMID 17011445
- [Background] Moon SH, Shin KH, Kim TH, Yoon M, Park S, Lee DH, Kim JW, Kim DW, Park SY, Cho KH. Dosimetric comparison of four different external beam partial breast irradiation techniques: three-dimensional conformal radiotherapy, intensity-modulated radiotherapy, helical tomotherapy, and proton beam therapy. Radiother Oncol. 2009 Jan;90(1):66-73. doi: 10.1016/j.radonc.2008.09.027. Epub 2008 Nov 5. PMID 18992950
- [Background] Kanai T, Kawachi K, Kumamoto Y, Ogawa H, Yamada T, Matsuzawa H, Inada T. Spot scanning system for proton radiotherapy. Med Phys. 1980 Jul-Aug;7(4):365-9. doi: 10.1118/1.594693. PMID 6248752
- [Background] Stanton AL, Krishnan L, Collins CA. Form or function? Part 1. Subjective cosmetic and functional correlates of quality of life in women treated with breast-conserving surgical procedures and radiotherapy. Cancer. 2001 Jun 15;91(12):2273-81. PMID 11413515
- [Background] Olivotto IA, Whelan TJ, Parpia S, Kim DH, Berrang T, Truong PT, Kong I, Cochrane B, Nichol A, Roy I, Germain I, Akra M, Reed M, Fyles A, Trotter T, Perera F, Beckham W, Levine MN, Julian JA. Interim cosmetic and toxicity results from RAPID: a randomized trial of accelerated partial breast irradiation using three-dimensional conformal external beam radiation therapy. J Clin Oncol. 2013 Nov 10;31(32):4038-45. doi: 10.1200/JCO.2013.50.5511. Epub 2013 Jul 8. PMID 23835717
- [Background] Julian, T.B., et al., Early Toxicity Results with 3-D Conformal External Beam Therapy (CEBT) from the NSABP B-39/RTOG 0413 Accelerated Partial Breast Irradiation (APBI) Trial. International Journal of Radiation Oncology • Biology • Physics. 81(2): p. S7.
- [Background] Vrieling C, Collette L, Fourquet A, Hoogenraad WJ, Horiot JC, Jager JJ, Pierart M, Poortmans PM, Struikmans H, Van der Hulst M, Van der Schueren E, Bartelink H. The influence of the boost in breast-conserving therapy on cosmetic outcome in the EORTC "boost versus no boost" trial. EORTC Radiotherapy and Breast Cancer Cooperative Groups. European Organization for Research and Treatment of Cancer. Int J Radiat Oncol Biol Phys. 1999 Oct 1;45(3):677-85. doi: 10.1016/s0360-3016(99)00211-4. PMID 10524422
- See also: Surveillance, Epidemiology and End Results Cancer Statistics Review — https://seer.cancer.gov/csr/1975_2014/